CLINICAL TRIAL: NCT04207437
Title: Daily Hand-Held Vibration Therapy for the Treatment of Chemotherapy Induced Peripheral Neuropathy (CIPN): A Pilot Study
Brief Title: Daily Hand-Held Vibration Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Erin Newton, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0677
Record Dates: First submitted 2019-12-11; First posted 2019-12-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Neuropathy; Cancer; Chemotherapeutic Drug - Induced Nephropathy; Chemotherapeutic Toxicity
Keywords: Neuropathy; Vibration
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be instructed to perform 3-minutes of vibration therapy per hand each day using a hand held vibration device for 4 weeks. The amount of time that subjects perform vibration therapy will be recorded on their Daily Compliance form and subjects will complete questionnaires daily and weekly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vibration Therapy (Experimental): Patients will hold a hand held vibrating device for 3 minutes on each hand daily for 4 weeks.
  Interventions: Device: Vibration therapy

INTERVENTIONS:
Device: Vibration therapy — vibration therapy using hand held vibration device

SUMMARY:
The purpose of this pilot study is to determine the safety and feasibility of a daily 3-minute hand-held vibration therapy intervention to reduce the severity of CIPN in the hands. The investigators hypothesize that daily vibration therapy can reduce the severity of patient's CIPN in their hands and improve CIPN-related quality of life. The hope is that results from this study will provide early data on the feasibility, efficacy, and most importantly, safety, of daily 3-minute hand-held vibration therapy needed to justify future clinical trials examining vibration therapy as a potential option for treating CIPN in the future.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older at enrollment
2. Able to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
3. Have completed chemotherapy ≥ 60 days prior to enrollment
4. Were exposed to neurotoxic chemotherapy with one or more of the following agents in the following doses: Paclitaxel (cumulative dose: ≥ 300 mg/m2) Docetaxel (cumulative dose: ≥ 100 mg/m2) Nab-paclitaxel (cumulative dose: ≥ 750 mg/m2) Oxaliplatin (cumulative dose: ≥ 510 mg/m2) Carboplatin (cumulative dose: ≥ 600 mg/m2) Cisplatin (cumulative dose: ≥ 200 mg/m2) Vincristine (cumulative dose: ≥ 4 mg/m2) Bortezomib (cumulative dose: ≥ 16 mg/m)
5. Continue to display evidence of sensory CIPN in the hands rated at a Grade ≥ 2 according the National Cancer Institute's Common Toxicity Criteria-Adverse Events (NCI-CTC-AE, Version 5.0) Scale ≥ 60 days post-chemotherapy
6. If solid tumor cancer, must have non-metastatic cancer
7. Agree to return to clinic for required study related measurements at specified intervals

Exclusion Criteria:

1. Have pre-existing neuropathy affecting the hands not related to chemotherapy (e.g., carpal tunnel syndrome, nerve compression, etc.)
2. Known diagnosis of diabetes mellitus.
3. Known contraindications for vibration therapy to hands, including deep venous thrombosis of the upper extremity or ongoing skin infection.
4. Will be receiving concurrent radiation of the upper-extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment- percentage of patients who agree to participate in the study after screening | recruitment period (up to 5 year after study starts)
Feasibility of compliance- percentage of vibration therapy sessions completed | 4 weeks
  Compliance with the daily vibration therapy sessions will be evaluated using data from a Daily Compliance Form Researchers will calculate the percentage of sessions that were completed calculated for each participant, on each hand. Participant compliance with the intervention will be considered acceptable if participants complete ≥ 80% of the sessions they were assigned.
Acceptability of Intervention- percentage of patients who answer agree on acceptability form | 4 weeks
  percentage of participants who answer "somewhat agree," "agree," or "strongly agree" on the intervention acceptability form
Change in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy twenty-item scale (CIPN20) scores | baseline, week 1, week 2, week 3, week 4
  CIPN 20 questionnaire scores will be compared to baseline weekly to identify an increase of 30% during the intervention period. The CIPN scores range from 20 to 80 with 80 being consistent with the most severe neuropathy symptoms

SECONDARY OUTCOMES:
Change in CIPN Severity via the CIPN20 questionnaire scores | baseline, weeks 1, 2, 3, and 4, 5, 6, 7, and week 8
  Summary statistics for the weekly CIPN-20 (n, mean, standard deviation, median, minimum, maximum)
Change in CIPN related Quality of Life via the Chemotherapy Induced Peripheral Neuropathy Quality of Life Scale | baseline, week 4, week 8
  Descriptive statistics (frequency and percentage for each category, mean and standard deviation of scores assigned to each category (range: 0-7)) will be used to describe the CIPN-related QOL participants have on each of the three categories related to quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Erin Newton, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health West, Avon, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Joe & Shelly Schwarz Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No